CLINICAL TRIAL: NCT07364474
Title: Evaluating Immune Response to Percutaneous Hepatic Perfusion With Melphalan for the Treatment of Ocular Melanoma Metastatic to the Liver
Brief Title: Immune Response to Percutaneous Hepatic Perfusion With Melphalan for Ocular Melanoma Metastatic to the Liver
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Eric Wehrenberg-Klee, MD, Dana-Farber/Harvard Cancer Center Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 25-679
Record Dates: First submitted 2025-12-16; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Uveal Melanoma
Keywords: Uveal Melanoma; Uveal Melanoma, Metastatic; Uveal Melanoma, Metastatic to liver
MeSH Terms: conditions — Uveal Melanoma; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Melphalan through Percutaneous Hepatic Perfusion (Other): Single arm
  Interventions: Drug: Melphalan through Percutaneous Hepatic Perfusion

INTERVENTIONS:
Drug: Melphalan through Percutaneous Hepatic Perfusion — Melphalan through Percutaneous Hepatic Perfusion will be received as standard of care,

SUMMARY:
This study seeks to better understand the liver's immune response to receiving chemotherapy agent melphalan through Percutaneous Hepatic Perfusion (PHP) for patients with Uveal Melanoma that has metastasized to the liver.

DETAILED DESCRIPTION:
Biopsies and blood samples will be collected before treatment to establish baseline measurements. Patients will then receive a single dose of Melphalan via Percutaneous Hepatic Perfusion (PHP) and return 21-28 days later for a follow-up biopsy and peripheral blood draw. Baseline and post-treatment samples will be compared to evaluate the immune response.

ELIGIBILITY:
Inclusion Criteria:

* Patient has histologically or cytologically confirmed diagnosis of uveal melanoma metastatic to the liver and is determined to be a candidate for percutaneous hepatic perfusion with melphalan
* The subject has read, signed and dated the Informed Consent Form (ICF), having been advised of the risks and benefits of the trial in a language understood by the subject.
* Age > 18 years at date of informed consent signature having the ability to comply with the protocol.
* Contrast-enhanced cross-sectional imaging of the abdomen (either CT or MRI) obtained within one month prior to study enrollment
* Measurable metastatic disease. Subject must have at least one site of metastatic disease ≥ 1 cm in size and amenable to percutaneous image-guided biopsy
* Life expectancy > 12 weeks.
* ECOG Performance Status of 0 or 1
* Laboratory requirements:
* ANC > 1 x 109/L
* Platelets > 75 x 109/L
* ALT / AST < 5 x ULN
* Total bilirubin <3 mg/dL
* INR <1.7
* GFR >30 ml/min

Exclusion Criteria:

* Lesion to undergo biopsy cannot have undergone prior radiation therapy or other locoregional therapy
* Continued adverse events from a previously administered chemotherapeutic agents. Grade 1 adverse events and ongoing toxicities such as alopecia are exempt
* Treatment with systemic corticosteroids exceeding the equivalent of 10 mg/day of prednisone or other systemic immunosuppressive medications (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, and anti-tumor necrosis factor [anti-TNF] agents) within 2 weeks prior to Day 1, or anticipated requirement for systemic immunosuppressive medications exceeding the equivalent of 10 mg/day of prednisone during the trial
* Patients who receive acute, low-dose, systemic corticosteroid medications (e.g., a one-time dose of dexamethasone for nausea) or for prevention of hypersensitivity reactions to contrast agents may be enrolled in the trial.
* Anticoagulant or anti-platelet medication that cannot be interrupted prior to biopsy
* Pregnant or lactating
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicated the use of an investigational drug or that could affect the interpretation of the results or render the patient at high risk from treatment complications.
* Treatment with systemic immunostimulatory agents (including but not limited to IFNs, interleukin [IL]-2) within 6 weeks or five half- lives of the drug, whichever was shorter, prior to Day 1.
* Treatment with immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies, anti-LAG-3 antibodies, within the past three months. Prior treatment with tebentafusp is allowed with no washout period required.
* Treatment with any investigational systemic medication within at least one month prior to biopsy. If an investigational agent is an immune checkpoint inhibitor, a three-month washout is required.
* Signs or symptoms clinically significant of infection within 2 weeks prior to Day 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Intratumoral CXCL13⁺ CD8⁺ T-cell infiltration following Percutaneous Hepatic Perfusion (PHP) | 3-4 weeks post treatment
  Change in the percentage of CXCL13⁺ CD8⁺ T cells in tumor biopsies between Day 0 (pre-treatment) and Day 28-42 (approximately 3-4 weeks post-treatment), as measured by single-cell RNA sequencing.

SECONDARY OUTCOMES:
Antigen-presenting cell (APC) populations and their activation state in the tumor microenvironment. | 28-42 day tumor biopsies
  Comparison of proportions and activation markers of dendritic cells and other APC subsets in pre-treatment (Day 0) and post-treatment (Day 28-42) tumor biopsies.
T-cell infiltration in tumor and adjacent hepatic parenchyma. | 28-42 days post treatment
  Change in FOXP3⁺ regulatory T-cell infiltration between pre-treatment (Day 0) and post-treatment (Day 28-42) tumor and parenchymal biopsies.
Single-cell RNA sequencing derived frequency of macrophages and myeloid-derived suppressor cells (MDSCs) | 28-42 days post treatment
  Change in the frequency of macrophages and myeloid-derived suppressor cells (MDSCs) between pre-treatment (Day 0) and post-treatment (Day 28-42) samples as assessed by single-cell RNA sequencing.
Single-cell RNA sequencing derived phenotype of macrophages and myeloid-derived suppressor cells (MDSCs) | 28-42 days post treatment
  Change in the phenotype of macrophages and myeloid-derived suppressor cells (MDSCs) between pre-treatment (Day 0) and post-treatment (Day 28-42) samples.
Immune cell populations with molecular and biochemical features of tissue and peripheral blood. | 28-42 days post treatment.
  Correlation between tissue-based immune cell changes and peripheral biomarkers (e.g. cytokine expression (ng/ml), ctDNA (mtm/ml)) assessed at Day 0 and Day 28-42, and with hepatic radiologic response assessed on CT/MRI as per clinical standard of care .

CONTACTS AND LOCATIONS:
Overall Officials: Eric Wehrenberg-Klee, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: alawless@mgb.org . The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication.
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu